CLINICAL TRIAL: NCT02376777
Title: Comparison of Accidents and Their Circumstances With Oral Anticoagulants. The CACAO Study
Brief Title: Comparison of Accidents and Their Circumstances With Oral Anticoagulants
Acronym: CACAO
Status: Completed | Type: Observational
Sponsor: CNGE IRMG Association (Other)
Collaborators: Floralis (Industry); University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: DCIC 15 09
Record Dates: First submitted 2015-02-26; First posted 2015-03-03 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Cardiovascular Complications; Hemorrhagic Disorders; Embolism and Thrombosis
Keywords: Anticoagulants; Antithrombins; Atrial Fibrillation; Intracranial haemorrhage; Gastrointestinal haemorrhage; Myocardial infarction; Stroke; Venous thrombosis; Primary care
MeSH Terms: conditions — Hemorrhagic Disorders; Embolism and Thrombosis; Atrial Fibrillation; Intracranial Hemorrhages; Gastrointestinal Hemorrhage; Myocardial Infarction; Stroke; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patient receiving NOAC: Follow up of patients receiving new oral anticoagulants (NOAC) medication
  Interventions: Other: Follow up
- Patient receiving VKA: Follow up of patients receiving vitamin K antagonist (VKA) medication
  Interventions: Other: Follow up

INTERVENTIONS:
Other: Follow up — each three months during one year of follow up, general practioners will entered health data in database (hemorrhagic events, changes of medication, biological data...)

SUMMARY:
Differences in efficacy and safety between new oral anticoagulants (NOAC) and vitamin K antagonist (VKA) in real practice remain uncertain.

The few existing ambulatory studies did not answer all NOAC specific issues, such as prescription habits and motives, patients characteristics, biological monitoring, as well as the occurrence of major and minor thromboembolic events, especially in France where warfarin is less frequently prescribed.

Therefore, in order to describe clinical and follow up characteristics of patients receiving oral anticoagulants, the investigators will set up a national prospective cohort to compare the occurrence of thromboembolic events between VKA and NOAC in primary care.

DETAILED DESCRIPTION:
The method includes the use of a national prospective observational cohort, involving 444 general practitioners From april to december 2014, health data of any adult patient consulting a general practitioner and receiving an oral anticoagulant treatment has been entered in a database. Each patient received an information for agreement to participate to the study (agreement for stastical analysis of their health data during one year follow up).

In March 2015, half of those patients will be chosen (stratification), using a matched stratification process, and will be followed up over one year. Every three months, data regarding the occurrence of therapeutics changes, episodes of excessive bleeding, and thromboembolic events will be collected by general practitioners.

The data will be analysed by: - describing the characteristics of patients receiving oral anticoagulant treatment; - describing the changes of medications over the year ; - comparing the occurrence of episodes of excessive bleeding ; - comparing the occurrence of thromboembolic events in patients using VKA versus patients using NOAC.

ELIGIBILITY:
Inclusion Criteria :

* Patient consulting a GP
* Patient Whatever the reason for consultation
* Aged >18 years
* Receiving oral anticoagulant treatment by NOAC (apixaban, dabigatran or rivaroxaban) or VKA (acenocoumarol, fluindione, or warfarin)
* Whatever the indication (prevention or treatment).
* Having the following indications for anticoagulant treatment : non-valvular atrial fibrillation, prevention of DVT / PE (excluding orthopedic post-surgery) treatment DVT / PE

Exclusion Criteria :

* Aged <18 years
* Receiving concomitant injectable anticoagulant treatment (including relay phase)
* Follow up impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with anticoagulant medication consulting their general practitioner will be included (N=7846), and after stratification, 4162 patients will be followed
Sampling Method: Probability Sample
Enrollment: 4162 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Clinical characteristics | at baseline
  The profile of patients receiving VKA or NOAC will be described by the following variables:
  * Molecule, duration, dosage
  * Indication: Atrial fibrillaton valvular or not / DVT / PE / Other, Prevention / Treatment
  * Age, sex, weight, height
  * Medication adherence ( as perceived by the GP )
  * Renal function
  * CHA2DS2-VASc Score
  * HAS-BLED Score
  * RIETE score
  * unstable INR
  * Comorbidities: anemia, diabetes, kidney disease, liver disease, hypertension, heart failure, stroke, peripheral vascular desease, myocardial infarction (MI).
  * Concomitant treatments: NSAIDs, antiplatelets, other treatments with potentials interactions

SECONDARY OUTCOMES:
Bleeding events | at baseline, 3, 6, 9 and 12 months
  Compare annual impact of bleeding events between patients receiving NOAC and VKA. Bleeding will be collected according to the International Society on Thrombosis and Haemostasis (ISTH) and BARC classification
Thrombotic events | at baseline, 3, 6, 9 and 12 months
  Compare annual impact of thrombotic events (Ischemic stroke, DVT, PE, acute coronary syndrome) between patients receiving NOAC and VKA on further indications : non-valvular ACFA (excluding mitral regurgitation grade 3 and 4), preventing DVT / PE , DVT/ EP treatment
Death | at baseline, 3, 6, 9 and 12 months
  Describe the causes of death (including EP or cardiac events)
Therapeutic classes | at baseline, 3, 6, 9 and 12 months
  Describe the changes of therapeutic classes and reasons in NOAC and VKA treated population. Changes in indication for medicines, changes in mode and type of anticoagulant therapy
Bleeding score | at baseline, 3, 6, 9 and 12 months
  Assess the relevance of different scores to predict the risk of bleeding. Comparison of the diagnostic performance of different classical scores by studying the corresponding AUC ROC curves

CONTACTS AND LOCATIONS:
Overall Officials: Joël COGNEAU, MD, Principal Investigator — IRMG; Paul FRAPPE, MD, Study Director — University of Saint-Etienne; Jean-Pierre JACQUET, MD, Study Director — University of Grenoble; Jean-Luc BOSSON, MD PhD, Study Director — University of Grenoble; François Lacoin, MD, Study Director — IRMG
Locations (33):
- France (33):
  - Office-based practitioner, Albens
  - Office-based practitioner, Bordeaux
  - Office-based practitioner, Chablis
  - Office-based general practitioner, Dessenheim
  - Office-based general practitioner, Dijon
  - Office-based practitioner, Flumet
  - Office-based practitioner, Gémenos
  - Office-based general practitioner, Grenay
  - Office-based general practitioner, Guesnain
  - Office-based general practitioner, Hatten
  - Office-based practitioner, Hinx
  - Office-based practitioner, La Madeleine
  - Office-based practitioner, Les Marches
  - Office-based practitioner, Limoges
  - Office-based practitioner, Mulsanne
  - Office-based practitioner, Outreau
  - Office-based general practitioner, Paris
  - Office-based general practitioner, Rupt-sur-Moselle
  - Office-based general practitioner, Saint-Amant-Tallende
  - Office-based practitioner, Saint-Etienne
  - Office-based practitioner, Saint-Georges-dOrques
  - Office-based practitioner, Saint-Jean-d'Arvey
  - Office-based practitioner, Saint-Jean-de-Braye
  - Office-based practitioner, Saultain
  - Office-based general practitioner, Sellières
  - Office-based practitioner, Seraincourt
  - Office-based general practitioner, Soisy-sous-Montmorency
  - Office-based general practioner, Strasbourg
  - Office-based practitioner, Tournus
  - Office-based general practitioner, Tours
  - Office-based practitioner, Villeurbanne
  - Office-based practitioner, Vitry-sur-Seine
  - Office-based general practitioner, Vourey

REFERENCES:
- [Background] Kearon C. Natural history of venous thromboembolism. Circulation. 2003 Jun 17;107(23 Suppl 1):I22-30. doi: 10.1161/01.CIR.0000078464.82671.78. PMID 12814982
- [Background] You JJ, Singer DE, Howard PA, Lane DA, Eckman MH, Fang MC, Hylek EM, Schulman S, Go AS, Hughes M, Spencer FA, Manning WJ, Halperin JL, Lip GYH. Antithrombotic therapy for atrial fibrillation: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e531S-e575S. doi: 10.1378/chest.11-2304. PMID 22315271
- [Background] Mantilla CB, Horlocker TT, Schroeder DR, Berry DJ, Brown DL. Frequency of myocardial infarction, pulmonary embolism, deep venous thrombosis, and death following primary hip or knee arthroplasty. Anesthesiology. 2002 May;96(5):1140-6. doi: 10.1097/00000542-200205000-00017. PMID 11981154
- [Background] Galanaud JP, Sevestre-Pietri MA, Bosson JL, Laroche JP, Righini M, Brisot D, Boge G, van Kien AK, Gattolliat O, Bettarel-Binon C, Gris JC, Genty C, Quere I; OPTIMEV-SFMV Investigators. Comparative study on risk factors and early outcome of symptomatic distal versus proximal deep vein thrombosis: results from the OPTIMEV study. Thromb Haemost. 2009 Sep;102(3):493-500. doi: 10.1160/TH09-01-0053. PMID 19718469
- [Background] Douketis J, Tosetto A, Marcucci M, Baglin T, Cosmi B, Cushman M, Kyrle P, Poli D, Tait RC, Iorio A. Risk of recurrence after venous thromboembolism in men and women: patient level meta-analysis. BMJ. 2011 Feb 24;342:d813. doi: 10.1136/bmj.d813. PMID 21349898
- [Background] Ruff CT, Giugliano RP, Braunwald E, Hoffman EB, Deenadayalu N, Ezekowitz MD, Camm AJ, Weitz JI, Lewis BS, Parkhomenko A, Yamashita T, Antman EM. Comparison of the efficacy and safety of new oral anticoagulants with warfarin in patients with atrial fibrillation: a meta-analysis of randomised trials. Lancet. 2014 Mar 15;383(9921):955-62. doi: 10.1016/S0140-6736(13)62343-0. Epub 2013 Dec 4. PMID 24315724
- [Background] Miller CS, Grandi SM, Shimony A, Filion KB, Eisenberg MJ. Meta-analysis of efficacy and safety of new oral anticoagulants (dabigatran, rivaroxaban, apixaban) versus warfarin in patients with atrial fibrillation. Am J Cardiol. 2012 Aug 1;110(3):453-60. doi: 10.1016/j.amjcard.2012.03.049. Epub 2012 Apr 24. PMID 22537354
- [Background] Adam SS, McDuffie JR, Ortel TL, Williams JW Jr. Comparative effectiveness of warfarin and new oral anticoagulants for the management of atrial fibrillation and venous thromboembolism: a systematic review. Ann Intern Med. 2012 Dec 4;157(11):796-807. doi: 10.7326/0003-4819-157-10-201211200-00532. PMID 22928173
- [Background] Uchino K, Hernandez AV. Dabigatran association with higher risk of acute coronary events: meta-analysis of noninferiority randomized controlled trials. Arch Intern Med. 2012 Mar 12;172(5):397-402. doi: 10.1001/archinternmed.2011.1666. Epub 2012 Jan 9. PMID 22231617
- [Background] Larsen TB, Rasmussen LH, Skjoth F, Due KM, Callreus T, Rosenzweig M, Lip GY. Efficacy and safety of dabigatran etexilate and warfarin in "real-world" patients with atrial fibrillation: a prospective nationwide cohort study. J Am Coll Cardiol. 2013 Jun 4;61(22):2264-73. doi: 10.1016/j.jacc.2013.03.020. Epub 2013 Apr 3. PMID 23562920
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Derived] Gaboreau Y, Frappe P, Vermorel C, Foote A, Bosson JL, Pernod G; CACAO study investigators. Oral anticoagulant safety in family practice: prognostic accuracy of Bleeding Risk Scores (from the CACAO study). Fam Pract. 2024 Feb 28;41(1):9-17. doi: 10.1093/fampra/cmad121. PMID 38281089
- [Derived] Frappe P, Cogneau J, Gaboreau Y, Abenhaim N, Bayen M, Guichard C, Jacquet JP, Lacoin F, Liebart S, Bertoletti L, Bosson JL; CACAO study investigators. Anticoagulants' Safety and Effectiveness in General Practice: A Nationwide Prospective Cohort Study. Ann Fam Med. 2020 Mar;18(2):131-138. doi: 10.1370/afm.2495. PMID 32152017
- [Derived] Frappe P, Cogneau J, Gaboreau Y, Abenhaim N, Bayen M, Calafiore M, Guichard C, Jacquet JP, Lacoin F, Bertoletti L; CACAO study investigators. Areas of improvement in anticoagulant safety. Data from the CACAO study, a cohort in general practice. PLoS One. 2017 Apr 6;12(4):e0175167. doi: 10.1371/journal.pone.0175167. eCollection 2017. PMID 28384199